CLINICAL TRIAL: NCT00003906
Title: Study of Tamoxifen and Raloxifene (STAR) for the Prevention of Breast Cancer
Brief Title: Study of Tamoxifen and Raloxifene (STAR) for the Prevention of Breast Cancer in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eli Lilly and Company (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NSABP P-2; CDR0000067081
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Raloxifene Hydrochloride; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Tamoxifen and placebo
  Interventions: Drug: Tamoxifen
- Group 2 (Experimental): Raloxifene and Placebo
  Interventions: Drug: Raloxifene

INTERVENTIONS:
Drug: Raloxifene — 60 mg/day plus placebo for 5 years
  Arms: Group 2
Drug: Tamoxifen — 20 mg/day plus placebo for 5 years
  Arms: Group 1

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using raloxifene and tamoxifen may fight breast cancer by blocking the uptake of estrogen by the tumor cells.

PURPOSE: Randomized double-blinded clinical trial to compare the effectiveness of raloxifene with that of tamoxifen in preventing breast cancer in postmenopausal women.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether raloxifene is more or less effective than tamoxifen in significantly reducing the incidence rate of invasive breast cancer in postmenopausal women.
* Evaluate the effects of tamoxifen and raloxifene on the incidence of intraductal carcinoma in situ, lobular carcinoma in situ, endometrial cancer, ischemic heart disease, fractures of the hip and spine, or Colles' fractures of the wrist in these participants.
* Evaluate the toxic effects of these regimens in these participants.
* Determine the effect of these regimens on the quality of life of these participants (at selected centers). (Quality of life evaluation closed to accrual effective 5/31/01.)

OUTLINE: This is a randomized, double-blind study. Participants are stratified by age (35 to 49 vs 50 to 59 vs over 59), race (black vs white vs other), history of lobular carcinoma in situ (yes vs no), prior hysterectomy (yes vs no), and estimated absolute risk of invasive breast cancer within 5 years (using the Gail model)(less than 2.0 vs 2.0-2.9 vs 3.0-4.9 vs 5.0 or greater). Participants are randomized to 1 of 2 arms.

* Arm I: Participants receive oral tamoxifen plus placebo daily for 5 years.
* Arm II: Participants receive oral raloxifene plus placebo daily for 5 years. Quality of life is assessed (at selected centers) at baseline and at 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, and 72 months. (Quality of life evaluation closed to accrual effective 5/31/01.)

Participants are followed annually after 5 years.

PROJECTED ACCRUAL: Approximately 19,000 participants will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Postmenopausal women at increased risk for developing invasive breast cancer, who meet one of the following criteria:

  * At least 12 months since spontaneous menstrual bleeding
  * Prior documented hysterectomy and bilateral salpingo-oophorectomy
  * At least 55 years of age with prior hysterectomy with or without oophorectomy
  * Age 35 to 54 with a prior hysterectomy without oophorectomy OR with a status of ovaries unknown with documented follicle-stimulating hormone level demonstrating elevation in postmenopausal range
* Histologically confirmed lobular carcinoma in situ treated by local excision only OR a minimum projected 5 year probability of invasive breast cancer of at least 1.66%, using Breast Cancer Risk Assessment Profile
* No clinical evidence of malignancy on physical exam within the past 180 days
* No evidence of suspicious or malignant disease on bilateral mammogram within the past year
* No bilateral or unilateral prophylactic mastectomy
* No prior invasive breast cancer or intraductal carcinoma in situ
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 35 and over

Sex:

* Female

Menopausal status:

* See Disease Characteristics

Performance status:

* No restricted normal activity for a significant portion of each day

Life expectancy:

* At least 10 years

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Complete blood count and differential normal
* Platelet count normal

Hepatic:

* SGOT or SGPT normal
* Bilirubin normal
* Alkaline phosphatase normal

Renal:

* Creatinine normal

Cardiovascular:

* No cerebral vascular accident, transient ischemic attack, atrial fibrillation, or uncontrolled hypertension
* No deep vein thrombosis

Pulmonary:

* No pulmonary embolus

Other:

* No other prior malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No concurrent nonmalignant disease that would preclude administration of tamoxifen or raloxifene
* No clinical depression, psychiatric condition, or addictive disorder
* No uncontrolled diabetes

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* At least 3 months since prior estrogen or progesterone replacement therapy, oral contraceptives, androgens, luteinizing hormone-releasing hormone analogs, prolactin inhibitors, or antiandrogens
* At least 3 months since prior tamoxifen, raloxifene, or other selective estrogen-receptor modulators of less than 3 months duration
* Concurrent Estring allowed

Radiotherapy:

* No prior breast radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No prior systemic adjuvant therapy for breast cancer
* No other participation in a cancer prevention or osteoporosis prevention study involving pharmacologic intervention(s)

  * NSABP-P-1 patients who received placebo are eligible
* No concurrent warfarin or cholestyramine
* Concurrent calcitonin or nonhormonal medication (e.g., cholecalciferol, fluoride, or bisphosphonates) allowed

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19747 (Actual)
Dates: Start 1999-05; Primary Completion 2005-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Incidence of invasive breast cancer; superiority of one of the therapies. | Time from randomization to the occurance of invasive breast cancer.
  Determine which of the following is true:
  1. compared to tamoxifen, raloxifene significantly reduces the incidence rate of invasive breast cancer;
  2. compared to raloxifene, tamoxifen significantly reduces the incidence rate of invasive breast cancer; or
  3. the statistical superiority of one of the treatments cannot be demonstrated and the choice of therapy should be based on benefit/risk considerations.

SECONDARY OUTCOMES:
Effect of the study therapies on the incidence of intraductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS). | Time from randomization to the occurance of DCIS or LCIS.
Effect of the study therapies on the incidence of endometrial cancer. | Time from randomization to the occurance of endometrial cancer.
Effect of the study therapies on the incidence of ischemic heart disease. | Time from randomization to the occurance of ischimic heart disease.
Effect of the study therapies on the incidence of fractures of the hip, spine, or Colles' fractures of the wrist. | Time from randomization to the occurance of fractures of the hip, spine, or Colles' fractures of the wrist.
Effect of the study therapies on the toxicity and side effects of each therapy. | Incidences of protocol defined toxicities and side effects.
Effect of the study therapies on participants' quality of life. | pre-entry, every 6 months for 5 years, and then annual after 5 years following randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Study Chair — NSABP Foundation Inc
Locations (516):
- United States (492):
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Breast Associates, Fayetteville, Arkansas
  - Surgical Associates, Fort Smith, Arkansas
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Medical Center - Anaheim/Orange County, Anaheim, California
  - Kaiser Permanente Medical Center - Baldwin Park, Baldwin Park, California
  - Kaiser Permanente Medical Center - Bellflower, Bellflower, California
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mills-Peninsula Health Services, Burlingame, California
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - Mount Diablo Medical Center, Concord, California
  - Corona Regional Medical Center, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Scripps Memorial Hospitals-Stevens Cancer Center - Encinitas, Encinitas, California
  - North Bay Cancer Center, Fairfield, California
  - Kaiser Permanente Medical Center - Fontana, Fontana, California
  - Crosson Cancer Center at St. Jude Medical Center, Fullerton, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Oncology/Hematology Associates, Granada Hills, California
  - Marin General Hospital Cancer Institute, Greenbrae, California
  - Kaiser Permanente Medical Center - Harbor City, Harbor City, California
  - Hemet Valley Medical Center, Hemet, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Valley Tumor Medical Group, Lancaster, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Todd Cancer Institute at Long Beach Memorial Medical Center, Long Beach, California
  - Pacific Shores Medical Group Comprehensive Hematology-Oncology Services - Long Beach, Long Beach, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Cecilia Gonzalez De La Hoya Cancer Center at White Memorial Medical Center, Los Angeles, California
  - Kaiser Foundation Hospital - West Los Angeles, Los Angeles, California
  - St. Vincent Medical Center - Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Mission Cancer Center at Mission Hospital, Mission Viejo, California
  - Sutter Gould Medical Foundation, Modesto, California
  - Leavey Cancer Center at Northridge Hospital Medical Center, Northridge, California
  - Breast Health Center, Oceanside, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - Ventura Hematology - Oncology Specialists - Oxnard, Oxnard, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Kaiser Permanente Medical Group, Panorama City, California
  - Huntington Cancer Center at Huntington Hospital, Pasadena, California
  - Wilshire Oncology Medical Group, Incorporated - Pomona, Pomona, California
  - North Valley Breast Clinic, Redding, California
  - Kaiser Permanente Medical Center - Riverside, Riverside, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Breast Cancer Group, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Torrance Memorial Medical Center, Torrance, California
  - Santa Clarita Valley Cancer Center - UCLA, Valencia, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Cener - Woodland Hills, Woodland Hills, California
  - Penrose Cancer Center, Colorado Springs, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - University of Connecticut Comprehensive Cancer Center at University of Connecticut Health Center, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - New Britain General Hospital, New Britain, Connecticut
  - Hospital of St. Raphael, New Haven, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Lawrence and Memorial Hospital, New London, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Hematology Oncology, P.C., Stamford, Connecticut
  - Northwestern Connecticut Oncology-Hematology Associates, Torrington, Connecticut
  - Windham Community Memorial Hospital, Williamantic, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Providence Hospital, Washington D.C., District of Columbia
  - JFK Medical Center, Atlantis, Florida
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Watson Clinic, Lakeland, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Medical Center, Orlando, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - West Florida Regional Medical Center, Pensacola, Florida
  - Cancer Research Network Inc., Plantation, Florida
  - Clinical Research Center of South Florida, Stuart, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Care and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush Copley Medical Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Rush Cancer Institute at Rush University Medical Center, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Our Lady of the Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - St. Francis Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Evanston Northwestern Health Care - Highland Park Hospital, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology Hematology Associates, Limited - Joliet, Joliet, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Mid-Illinois Hematology-Oncology Associates, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute, Olympia Fields, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Trinity Medical Center - West, Rock Island, Illinois
  - Rockford Clinic, Rockford, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Edward H. Kaplan MD and Associates, Skokie, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana Community Cancer Care, Incorporated, Indianapolis, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Indiana Regional Cancer Center, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Oncology Institute of Greater Lafayette, Lafayette, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Ball Memorial Hospital Cancer Center, Muncie, Indiana
  - Community Hospital, Munster, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - Medical Associates, Clinton, Iowa
  - Jennie Edmundson Memorial Hospital, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - Cedar Valley Medical Specialists, P.C., Waterloo, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - King's Daughters Medical Center, Ashland, Kentucky
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - HCA Kings Daughters Memorial Hospital, Frankfort, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Norton Healthcare Cancer Center, Louisville, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Ochsner Clinic of Baton Rouge, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Cancer Care Specialists, Houma, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Cancer Treatment Center at Christus Schumpert St. Mary Place, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Goodall Hospital, Sanford, Maine
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Harvard Vanguard Medical Associates - Kenmore, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Caritas Norwood Hospital, Norfolk, Massachusetts
  - NSMC Cancer Center, Peabody, Massachusetts
  - Berkshire Physicians and Surgeons, P.C., Pittsfield, Massachusetts
  - Jordan Hospital Club Cancer Center, Plymouth, Massachusetts
  - Baystate Regional Cancer Program at Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System, Battle Creek, Michigan
  - Bay Diagnostic Center for Women, Bay City, Michigan
  - Community Health Center of Branch County, Coldwater, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Flint Hematology Oncology, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Center for Hematology/Oncology, Jackson, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Michigan State University Department of Surgery, Lansing, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - Mercy Memorial Hospital, Corporation, Monroe, Michigan
  - Community Cancer Care Specialist, Mount Clemens, Michigan
  - Memorial Healthcare, Owosso, Michigan
  - Blue Water Oncology PC, Port Huron, Port Huron, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Saint Mary's Seton Cancer Institute, Saginaw, Michigan
  - Providence Cancer Institute at Providence Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - St. Luke's Medical Clinic, Duluth, Minnesota
  - Minnesota Cooperative Group Program, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Coast Oncology/Hematology, P.L.L.C., Biloxi, Mississippi
  - Mid Delta Family Practice, Cleveland, Mississippi
  - Hattiesburg Clinic, P.A., Hattiesburg, Mississippi
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - North Mississippi Hematology and Oncology Associates, Limited, Tupelo, Mississippi
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Missouri Cancer Care, P.C. - St. Charles, Saint Charles, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Midwest Hematology Oncology Group, Inc., St Louis, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - Ozarks Medical Center, West Plains, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Montana Cancer Institute - Benefis Healthcare, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Francis Medical Center, Grand Island, Nebraska
  - Cancer Center at the Good Samaritan Health Systems, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - Alegent Health - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Southern New Hampshire Medical Center, Nashua, New Hampshire
  - Cooper Cancer Institute, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Warren Hospital, Phillipsburg, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Capital Health System at Mercer, Trenton, New Jersey
  - Underwood Memorial Hospital, Woodbury, New Jersey
  - Hematology-Oncology Associates, PC, Albuquerque, New Mexico
  - Lovelace Medical Center at Lovelace Sandia Health System, Albuquerque, New Mexico
  - New Mexico Oncology-Hematology Consultants, Limited, Albuquerque, New Mexico
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, P.C. - Albany Regional Cancer Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Louis Busch Hager Cancer Center at Mary Imogene Bassett Hospital, Cooperstown, New York
  - Charles R. Wood Foundation Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - New York Oncology Hematology, P.C. - Latham, Latham, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Saint Vincent Catholic Medical Center of New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - St. Francis Hospital and Health Centers, Poughkeepsie, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Genesee Surgical Associates, Rochester, New York
  - Gynecologic Oncology Associates, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - University Hospital - Stony Brook, Stony Brook, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - Comprehensive Cancer Center at Our Lady of Mercy Medical Center, The Bronx, New York
  - Mission Hospitals, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Gaston Hematology and Oncology, Gastonia, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Leo W. Jenkins Cancer Center of University Health Systems of Eastern Carolina, Greenville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Cornerstone Surgery, High Point, North Carolina
  - Raleigh Hematology/Oncology Associates, P.A. - Rex Cancer Center, Raleigh, North Carolina
  - Cancer Center at Iredell Memorial Hospital, Statesville, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Quain & Ramstad Clinic, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Cancer Center at Christ Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Fairview Hospital, Cleveland, Ohio
  - Kaiser Permanente, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - Flower Hospital - ProMedica Health System, Sylvania, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - St. Charles Hospital, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated, Toledo, Ohio
  - Cleveland Clinic Health System STAR BCPT, Warrensville Heights, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Muskogee Regional Medical Center, Muskogee, Oklahoma
  - Frank C. Love Cancer Institute at St. Anthony Hospital, Oklahoma City, Oklahoma
  - Central Oklahoma Cancer Center at INTEGRIS Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Health Center, Oklahoma City, Oklahoma
  - Oklahoma University Medical Center at University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - St. Charles Medical Center, Bend, Oregon
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Sacred Heart Hospital, Allentown, Pennsylvania
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - Bon Secours-Holy Family Health System, Altoona, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Community Hopital, Ephrata, Pennsylvania
  - Regional Cancer Center - Erie, Erie, Pennsylvania
  - Pinnacle Health Regional Cancer Center at Pinnacle Health System, Harrisburg, Pennsylvania
  - Mercy Community Hospital, Havertown, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Saint Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Cancer Center at Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Frankford Hospital, Philadelphia, Pennsylvania
  - Chestnut Hill Healthcare, Philadelphia, Pennsylvania
  - Fox Chase - Temple Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Mercy Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Crozer-Chester Medical Center, Upland, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Wellspan Health - York Cancer Center, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Roper St. Francis Healthcare - Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Richland Memorial Hospital, Columbia, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - U.T. Cancer Institute at University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Cancer Institute - Memphis at Baptist Memorial Hospital - Memphis, Memphis, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Hendrick Cancer Center, Abilene, Texas
  - Harrington Cancer Center, Amarillo, Texas
  - Julie and Ben Rogers Cancer Center, Beaumont, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Charles A. Sammons Cancer Center, Dallas, Texas
  - Methodist Dallas Medical Center, Dallas, Texas
  - Providence Memorial Hospital, El Paso, Texas
  - Harris Methodist Fort Worth, Fort Worth, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Baylor Medical Center at Garland, Irving, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Sanchez Cancer Center, Laredo, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Southwest Cancer and Research Center at University Medical Center, Lubbock, Texas
  - Memorial Health System of East Texas, Lufkin, Texas
  - Baylor/Richardson Cancer Center, Richardson, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Mountainview Medical, Berlin Corners, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Community Cancer Center at Rutland Regional Medical Center, Rutland, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Cancer Center of the Piedmont, Inc., Danville, Virginia
  - Danville Hematology and Oncology, Incorporated, Danville, Virginia
  - Virginia Oncology Associates - Newport News, Newport News, Virginia
  - Henrico Doctors' Hospital - Parham Campus, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Flynn Cancer Center at Providence Everett Medical Center - Pacific Campus, Everett, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Cancer Care Northwest - Spokane North, Spokane, Washington
  - Rockwood Clinic P.S., Spokane, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Yakima Regional Cancer Care Center, Yakima, Washington
  - David Lee Cancer Center at Charleston Area Medical Center, Charleston, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Oncology Alliance, S.C., Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - UW Cancer Center Wausau Hospital, Wausau, Wisconsin
- Canada (23):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - University Hospital - U.B.C. Site, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Familial Oncology Program, Kingston, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - North York General Hospital, Ontario, North York, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Care, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Women's College Ambulatory Care Center, Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Ville Marie Breast Center, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - Hopital du Saint-Sacrement, Quebec, Québec, Quebec
  - Centre Universitaire de Sante de L'Estrie, Sherbrooke, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- MBCCOP - San Juan, San Juan, Puerto Rico

REFERENCES:
- [Background] Cronin WM, Cecchini RS, Wickerham DL, et al.: Factors associated with participant adherence in the NSABP Study of Tamoxifen and Raloxifene (STAR). [Abstract] J Clin Oncol 26 (Suppl 15): A-6518, 2008.
- [Background] Land SR, Ritter MW, Costantino JP, Julian TB, Cronin WM, Haile SR, Wolmark N, Ganz PA. Compliance with patient-reported outcomes in multicenter clinical trials: methodologic and practical approaches. J Clin Oncol. 2007 Nov 10;25(32):5113-20. doi: 10.1200/JCO.2007.12.1749. PMID 17991930
- [Background] Gradishar WJ, Cella D. Selective estrogen receptor modulators and prevention of invasive breast cancer. JAMA. 2006 Jun 21;295(23):2784-6. doi: 10.1001/jama.295.23.jed60037. Epub 2006 Jun 5. No abstract available. PMID 16754726
- [Result] Vogel VG. The NSABP Study of Tamoxifen and Raloxifene (STAR) trial. Expert Rev Anticancer Ther. 2009 Jan;9(1):51-60. doi: 10.1586/14737140.9.1.51. PMID 19105706
- [Result] Wickerham DL, Costantino JP, Vogel VG, Cronin WM, Cecchini RS, Ford LG, Wolmark N. The use of tamoxifen and raloxifene for the prevention of breast cancer. Recent Results Cancer Res. 2009;181:113-9. doi: 10.1007/978-3-540-69297-3_12. PMID 19213563
- [Result] Ganz PA, Land SR, Wickerham DL, et al.: The Study of Tamoxifen and Raloxifene (STAR): Change in patient-reported outcomes (PROs) after the end of treatment. [Abstract] J Clin Oncol 25 (Suppl 18): A-1506, 2007.
- [Result] Ganz PA, Land SR, Wickerham DL, et al.: The study of tamoxifen and raloxifene (STAR): first report of patient-reported outcomes (PROs) from the NSABP P-2 breast cancer prevention study. [Abstract] J Clin Oncol 24 (Suppl 18): A-LBA561, 2006.
- [Result] Land SR, Wickerham DL, Costantino JP, Ritter MW, Vogel VG, Lee M, Pajon ER, Wade JL 3rd, Dakhil S, Lockhart JB Jr, Wolmark N, Ganz PA. Patient-reported symptoms and quality of life during treatment with tamoxifen or raloxifene for breast cancer prevention: the NSABP Study of Tamoxifen and Raloxifene (STAR) P-2 trial. JAMA. 2006 Jun 21;295(23):2742-51. doi: 10.1001/jama.295.23.joc60075. Epub 2006 Jun 5. PMID 16754728
- [Result] Vogel VG, Costantino JP, Wickerham DL, et al.: The effects of tamoxifen versus raloxifene on the risk of developing noninvasive breast cancer in the NSABP study of tamoxifen and raloxifene (STAR) P-2 trial. [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-33, S16, 2006.
- [Result] Vogel VG, Costantino JP, Wickerham DL, Cronin WM, Cecchini RS, Atkins JN, Bevers TB, Fehrenbacher L, Pajon ER Jr, Wade JL 3rd, Robidoux A, Margolese RG, James J, Lippman SM, Runowicz CD, Ganz PA, Reis SE, McCaskill-Stevens W, Ford LG, Jordan VC, Wolmark N; National Surgical Adjuvant Breast and Bowel Project (NSABP). Effects of tamoxifen vs raloxifene on the risk of developing invasive breast cancer and other disease outcomes: the NSABP Study of Tamoxifen and Raloxifene (STAR) P-2 trial. JAMA. 2006 Jun 21;295(23):2727-41. doi: 10.1001/jama.295.23.joc60074. Epub 2006 Jun 5. PMID 16754727
- [Derived] McCaskill-Stevens W, Wilson JW, Cook ED, Edwards CL, Gibson RV, McElwain DL, Figueroa-Moseley CD, Paskett ED, Roberson NL, Wickerham DL, Wolmark N. National Surgical Adjuvant Breast and Bowel Project Study of Tamoxifen and Raloxifene trial: advancing the science of recruitment and breast cancer risk assessment in minority communities. Clin Trials. 2013 Apr;10(2):280-91. doi: 10.1177/1740774512470315. Epub 2013 Jan 18. PMID 23335675
- [Derived] Cecchini RS, Costantino JP, Cauley JA, Cronin WM, Wickerham DL, Land SR, Weissfeld JL, Wolmark N. Body mass index and the risk for developing invasive breast cancer among high-risk women in NSABP P-1 and STAR breast cancer prevention trials. Cancer Prev Res (Phila). 2012 Apr;5(4):583-92. doi: 10.1158/1940-6207.CAPR-11-0482. Epub 2012 Feb 7. PMID 22318751
- [Derived] Goetz MP, Schaid DJ, Wickerham DL, Safgren S, Mushiroda T, Kubo M, Batzler A, Costantino JP, Vogel VG, Paik S, Carlson EE, Flockhart DA, Wolmark N, Nakamura Y, Weinshilboum RM, Ingle JN, Ames MM. Evaluation of CYP2D6 and efficacy of tamoxifen and raloxifene in women treated for breast cancer chemoprevention: results from the NSABP P1 and P2 clinical trials. Clin Cancer Res. 2011 Nov 1;17(21):6944-51. doi: 10.1158/1078-0432.CCR-11-0860. Epub 2011 Aug 31. PMID 21880792
- [Derived] Vogel VG, Costantino JP, Wickerham DL, Cronin WM, Cecchini RS, Atkins JN, Bevers TB, Fehrenbacher L, Pajon ER, Wade JL 3rd, Robidoux A, Margolese RG, James J, Runowicz CD, Ganz PA, Reis SE, McCaskill-Stevens W, Ford LG, Jordan VC, Wolmark N; National Surgical Adjuvant Breast and Bowel Project. Update of the National Surgical Adjuvant Breast and Bowel Project Study of Tamoxifen and Raloxifene (STAR) P-2 Trial: Preventing breast cancer. Cancer Prev Res (Phila). 2010 Jun;3(6):696-706. doi: 10.1158/1940-6207.CAPR-10-0076. Epub 2010 Apr 19. PMID 20404000